CLINICAL TRIAL: NCT06062511
Title: Evaluation of Nutrikinetic and Bioavailability of Phenolic Compounds From ESIT12, a Poplar-type Propolis Dry Extract
Brief Title: Poplar-type Propolis Dry Extract ESIT12 : Nutrikinetic and Bioavailability Studies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fytexia (Industry)
Collaborators: Universidad Católica San Antonio de Murcia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: ESIT12BAS
Record Dates: First submitted 2023-09-07; First posted 2023-10-02 (Actual); Last update posted 2023-12-08 (Actual); Status verified 2023-12

CONDITIONS: Nutrition, Healthy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Verum ESIT12 D (Experimental): This arm receives 400 mg of ESIT12 and 150 mg of carriers from ESIT12
  Interventions: Dietary Supplement: ESIT12 D
- Verum ESIT12 4D (Experimental): This arm receives 1600 mg of ESIT12 and 600 mg of carriers from ESIT12
  Interventions: Dietary Supplement: ESIT12 4D
- Placebo (Placebo Comparator): This arm receives 550 mg of carriers from ESIT12
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: ESIT12 D — ESIT12 is a poplar-type propolis powder extract containing phenolic compounds from flavonoids and phenolic acids family. ESIT12 D contains 400 mg of ESIT12
  Arms: Verum ESIT12 D
Dietary Supplement: ESIT12 4D — ESIT12 is a poplar-type propolis powder extract containing phenolic compounds from flavonoids and phenolic acids family. ESIT12 4D contains 1600 mg of ESIT12
  Arms: Verum ESIT12 4D
Dietary Supplement: Placebo — Placebo is composed of the carriers of ESIT12 : arabic gum, sucrose and silicon dioxide mix
  Arms: Placebo

SUMMARY:
The aim of this study is to investigate phenolic compounds from ESIT12, a poplar-type propolis ingredient, bioavailability and nutrikinetics by measuring urinary excretion and metabolic profile over 48h by means of high-performance liquid chromatography coupled with tandem mass spectrometry (HPLC-MS/MS). The study follows a cross-over, double-blind, randomized and placebo control design on 10 healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form.
2. Stated willingness to comply with all study procedures and availability for the duration of the study.
3. Male and female with 40% min. and 60% max. of each sex.
4. Aged 25 to 69 years old
5. BMI range (18.5 - 29.99)
6. In good general health as evidenced by medical history
7. Ability to take oral supplementation and be willing to adhere to the regimen
8. Agreement to adhere to Lifestyle Considerations (controlled diet) throughout study duration

Exclusion Criteria:

1. Current use of any medication or food supplement
2. Antibiotic use less than 12 weeks before the study
3. Pregnancy or lactation
4. Known allergic reactions to components of the supplement, i.e., bee products (specially propolis) and known allergy (general)
5. Metabolic disorders or any kind of disease
6. Current smoker

Ages: 25 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Male and female with 40% min. and 60% max. of each sex.
Enrollment: 10 (Actual)
Dates: Start 2023-07-22 (Actual); Primary Completion 2023-10-10 (Actual); Study Completion 2023-10-10 (Actual)

PRIMARY OUTCOMES:
Change in plasma area under the curve (AUC) of phenolic metabolites after acute ingestion of the supplement/placebo | Baseline (pre-ingestion) to 24 hour post-ingestion
  Plasma samples will be collected in EDTA tubes in baseline before supplement/placebo intake (0h) and up to 24h according to the time frame. Phenolic compounds metabolites in plasma will be identified and quantified by HPLC-MS. Targeted metabolites are phenolic acids and flavonoids derivatives. For each identified and quantified metabolite the area under the curve (0-24 hour) in nmol/L-h is measured.
Change in plasma maximal concentration (Cmax) of phenolic metabolites after acute ingestion of the supplement/placebo | Baseline (pre-ingestion) and 0.5 hour, 1 hour, 2 hour, 3 hour, 4 hour, 6 hour, 8 hour, 10 hour, 24 hour post-ingestion
  Plasma samples will be collected in EDTA tubes in baseline before supplement/placebo intake (0h) and up to 24h according to the time frame. Phenolic compounds metabolites in plasma will be identified and quantified by HPLC-MS. Targeted metabolites are phenolic acids and flavonoids derivatives. For each identified and quantified metabolite the maximal concentration in nmol/L is measured.
Change in plasma time to reach maximal concentration (Tmax) of phenolic metabolites after acute ingestion of the supplement/placebo | Baseline (pre-ingestion) and 0.5 hour, 1 hour, 2 hour, 3 hour, 4 hour, 6 hour, 8 hour, 10 hour, 24 hour post-ingestion
  Plasma samples will be collected in EDTA tubes in baseline before supplement/placebo intake (0h) and up to 24h according to the time frame. Phenolic compounds metabolites in plasma will be identified and quantified by HPLC-MS. Targeted metabolites are phenolic acids and flavonoids derivatives. For each identified and quantified metabolite the time to reach maximum concentration in hour is measured.
Change in urine area under the curve (AUC) phenolic metabolites excretion after acute ingestion of the supplement/placebo | Baseline (pre-ingestion) to 48 hour post-ingestion
  Urine samples will be collected in baseline (0h pre-ingestion) and up to 48h according to the time frame. Phenolic compounds metabolites in urine will be identified and quantified by HPLC-MS. Targeted metabolites are phenolic acids and flavonoids derivatives. For each identified and quantified metabolite the area under the curve (0-24 hour) in nmol/L-h is measured.
Change in urine maximal concentration (Cmax) phenolic metabolites excretion after acute ingestion of the supplement/placebo | Baseline (pre-ingestion) and 0 hour - 3 hour, 3 hour - 6 hour, 6 hour - 10 hour, 10 hour - 14 hour, 14 hour - 24 hour, 24 hour - 36 hour and 36 hour - 48 hour post-ingestion
  Urine samples will be collected in baseline (0h pre-ingestion) and up to 48h according to the time frame. Phenolic compounds metabolites in urine will be identified and quantified by HPLC-MS. Targeted metabolites are phenolic acids and flavonoids derivatives. For each identified and quantified metabolite the maximal concentration in nmol/L is measured.
Change in urine time to reach maximal concentration (Tmax) phenolic metabolites excretion after acute ingestion of the supplement/placebo | Baseline (pre-ingestion) and 0 hour - 3 hour, 3 hour - 6 hour, 6 hour - 10 hour, 10 hour - 14 hour, 14 hour - 24 hour, 24 hour - 36 hour and 36 hour - 48 hour post-ingestion
  Urine samples will be collected in baseline (0h pre-ingestion) and up to 48h according to the time frame. Phenolic compounds metabolites in urine will be identified and quantified by HPLC-MS. Targeted metabolites are phenolic acids and flavonoids derivatives. For each identified and quantified metabolite the time to reach maximum concentration in hour is measured.

CONTACTS AND LOCATIONS:
Overall Officials: Pedro E. Alcaraz, PhD, Principal Investigator — UCAM
Locations (1):
- Universidad Católica San Antonio de Murcia, Guadalupe, Murcia, Spain

IPD SHARING:
Plan to Share IPD: No